CLINICAL TRIAL: NCT05784064
Title: Multicenter Survey About Acute Uncomplicated Diverticulitis Management
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fundación de Investigación Biomédica - Hospital Universitario de La Princesa (Other)
Responsible Party: Sponsor
Other Study IDs: 4489
Record Dates: First submitted 2023-03-13; First posted 2023-03-24 (Actual); Last update posted 2023-03-24 (Actual); Status verified 2023-03

CONDITIONS: Acute Uncomplicated Diverticulitis
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Survey — This is a nationalwide survey developed in order to know the management of patients diagnosed of acute uncomplicated diverticulitis.

SUMMARY:
Acute uncomplicated diverticulitis is a quite prevalent situation and consultation in the emergency department.

Its management has progresively changed towards a more conservative one and it is currently recommended in several guidelines the option of avoiding antibiotics in certain highly selected cases.

Nevertheless, the implantation of such recommendations in current clinical pratice is unknown and, hypothesizing it was still low, the reasons for such reluctancy are also unknown.

Both aspects can be considered quite interesting in order to design a specific plan in order to overcome such difficulties.

In order to do so, an online survery was designed and colorectal surgeons along Spain, based in the census of the Young Group from the Spanish Association of Colorectal Surgery were invited to participate. Invitations were distributed along usual communication channels of this group, such as email or chat mobile phone applications. All the responses to the survey will be analyzed in order to find out how many hospitals are using current managemente without antibiotics, its characteristics and, opposite, what are the main reasons for those hospitals that are not using it yet.

ELIGIBILITY:
Inclusion Criteria:

* Colorectal surgeons.
* Surgeons with emergency surgery activity.

Exclusion Criteria:

* Any other medical speciality.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Every surgeon with emergency surgery activity or colorectal surgeons that work at any Spanish hospital.
Sampling Method: Probability Sample
Enrollment: 56 (Estimated)
Dates: Start 2022-12-13 (Actual); Primary Completion 2023-04-10 (Estimated); Study Completion 2023-04-30 (Estimated)

PRIMARY OUTCOMES:
Acute uncomplicated diverticulitis management without antibiotics | 3rd january 2023-30th may 2023
  Rate of hospitals that includes management without antibiotics

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario de La Princesa, Madrid, Spain